CLINICAL TRIAL: NCT01410344
Title: Allogeneic Hematopoietic Cell Transplant for Hematological Cancers and Myelodysplastic Syndromes in HIV-Infected Individuals (BMT CTN #0903)
Brief Title: Allogeneic Transplant in HIV Patients (BMT CTN 0903)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Cancer Institute (NCI) (NIH); Blood and Marrow Transplant Clinical Trials Network (Network); National Marrow Donor Program (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMTCTN0903; U01HL069294 (NIH); BMT CTN 0903 (Other: Blood and Marrow Transplant Clinical Trials Network); 5U24CA076518 (NIH)
Record Dates: First submitted 2011-08-03; First posted 2011-08-05 (Estimated); Results first posted 2018-05-24 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Leukemia; Lymphoma; HIV
Keywords: HIV; ALL; AML; MDS; Non-Hodgkin Lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Lymphoma, Non-Hodgkin | interventions — fludarabine; Busulfan; fludarabine phosphate; Melphalan; Cyclophosphamide; Whole-Body Irradiation; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Allogeneic Transplant (Other): One regimen from either reduced-intensity conditioning (RIC) (Fludarabine and Busulfan; or Fludarabine and Melphalan) or myeloablative conditioning (MAC) (Busulfan and Fludarabine; or Cyclophosphamide and Total Body Irradiation) will be administered prior to allogeneic hematopoietic cell transplantation (HCT).
  Interventions: Drug: Fludarabine and Busulfan; Drug: Fludarabine and Melphalan; Drug: Busulfan and Fludarabine; Drug: Cyclophosphamide and Total Body Irradiation

INTERVENTIONS:
Drug: Fludarabine and Busulfan — RIC Regimen (Flu/Bu): Fludarabine total dose: 120-180 mg/m^2, Busulfan: ≤ 8 mg/kg PO or 6.4 mg/kg IV). Recommended regimen:
  * Days -6 to -2: Flu (30 mg/m^2/day, total dose of 150 mg/m^2)
  * Days -5 to -4: Busulfan (4mg/kg/day PO or 3.2 mg/kg IV, 130 mg/m^2/day, total dose of 8 mg/kg PO or 6.4 mg/kg IV, or 260 mg/m^2 IV, respectively)
  Patients with a creatinine clearance of 40-70 ml/min (measured or calculated) should have a 20 percent dose reduction in Fludarabine dosage.
  Busulfan will be dosed according to the recipient's ideal body weight (IBW), unless the patient weighs more than 125 percent of IBW, in which case the drug will be dosed according to the adjusted IBW.
  Other Names: Fludara and Busulfex
Drug: Fludarabine and Melphalan — RIC Regimen (Flu/Mel): Fludarabine total dose: 120-180 mg/m^2, Melphalan total dose: less than or equal to 150 mg/m^2. Recommended regimen:
  * Days -5 to -2: Flu (30mg/m^2/day, total dose of 120 mg/m^2)
  * Day -1: Mel (140mg/m^2)
  Patients with a creatinine clearance of 40-70 ml/min (measured or calculated) should have a 20 percent dose reduction in Fludarabine dosage.
  Other Names: Fludara and Alkeran
Drug: Busulfan and Fludarabine — MAC Regimen (Bu/Flu): Fludarabine total dose: 120-180mg/m^2 Busulfan total dose less than or equal to 16mg/kg PO or 12.8 mg/kg IV. Recommended regimen:
  * Days -5 to -2: Busulfan (4 mg/kg/day PO with Bu Css 900 plus/equal to 100 ng/mL (or per institutional standard), 3.2 mg/kg/day IV or 130 mg/m^2/day IV; total dose of 16 mg/kg, 12.8 mg/kg or 520 mg/m^2, respectively)
  * Days -5 to -2: Flu (30 mg/m^2/day, total dose of 120 mg/m^2)
  Patients with a creatinine clearance of 40-70 ml/min (measured or calculated) should have a 20 percent dose reduction in Fludarabine dosage.
  Busulfan will be dosed according to the recipient's ideal body weight (IBW), unless the patient weighs more than 125 percent of IBW, in which case the drug will be dosed according to the adjusted IBW.
  Other Names: Busulfex and Fludara
Drug: Cyclophosphamide and Total Body Irradiation — MAC Regimen (Cy/TBI): Cyclophosphamide total dose: 120 mg/kg, Fractionated TBI total dose: 1200-1420 cGy Recommended regimen:
  * Days -7 to -4: TBI (total dose of 1200-1420 cGy)
  * Days -3 to -2: Cy (60 mg/kg/day, total dose of 120 mg/kg)
  Cyclophosphamide will be dosed according to the recipient's ideal body weight (IBW), unless the patient weighs less than IBW, in which case the drug will be dosed according to the actual body weight.
  Other Names: Cytoxan® and radiation

SUMMARY:
The rationale for this trial is to demonstrate the feasibility and safety of allogeneic HCT for patients with chemotherapy-sensitive hematological malignancies and coincident HIV-infection. In particular, the trial will focus on the 100-day non-relapse mortality as an indicator of the safety of transplant in this patient population. Correlative assays will focus upon the incidence of infectious complications in this patient population, the evolution of HIV infection and immunological reconstitution. Where feasible (and when this can be accomplished without compromise of either the donor quality or the timeliness of transplantation), an attempt will be made to identify donors who are homozygotes for the delta32 mutation for CCR5.

DETAILED DESCRIPTION:
The study is designed to evaluate the feasibility and safety of reduced-intensity and fully-ablative allogeneic hematopoietic cell transplantation (HCT) for patients with hematological malignancies or myelodysplastic syndromes (MDS) who have HIV infection. The goal of the study is to assess the 100 day Non-relapse Mortality as well as immunological reconstitution in this patient population. Where feasible, an attempt will be made to identify human leukocyte antigen (HLA)-compatible hematopoietic stem cell donors who are homozygotes for the delta32 mutation of the chemokine receptor 5 (CCR5delta32). Patients will undergo a treatment plan review prior to registration on the trial. All patients will undergo allogeneic HCT from a matched sibling or unrelated donor.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infection, as documented by a rapid HIV test or any FDA-Approved HIV-1 Enzyme or Chemiluminescence Immunoassay (E/CIA) test kit and confirmed by Western Blot at any time prior to study entry. HIV antigen, plasma HIV-1 RNA, or a secondary antibody test by a method other than rapid HIV and E/CIA is acceptable as an alternative test. Alternatively, if a rapid HIV test or any FDA-Approved HIV-1 Enzyme or Chemiluminescence Immunoassay (E/CIA) test is not available, two HIV-1 RNA values ≥ 2000 copies/mL at least 24 hours apart performed by any laboratory that has CLIA certification, or its equivalent, may be used to document infection.
2. Patients must be willing to comply with effective Antiretroviral Therapy.
3. Patients must be ≥ 15 years of age.
4. Hematological malignancy associated with a poor prognosis with medical therapy alone. Diagnoses to be included:

   1. Patients with the diagnosis of Acute Myeloid or Lymphocytic Leukemia (AML or ALL) in first or second complete remission.
   2. Patients with advanced myelodysplastic syndromes (MDS), including those with International Prognostic Scoring System (IPSS) Int-2 and high-risk disease with less than 10% marrow blasts and no circulating myeloblasts after most recent therapy. Patients with acute leukemia that develops from a pre-existing MDS must meet the inclusion criteria for patients with AML detailed above.
   3. Hodgkin Lymphoma beyond first remission achieving at least a partial response to most recent therapy with no evidence of progression prior to transplant.
   4. Non-Hodgkin Lymphoma beyond first remission achieving at least a partial response to most recent therapy with no evidence of progression prior to transplant.
5. Donor/Recipient HLA Matching:

   1. Related donor: must be an 8/8 match at HLA-A, -B, -C, (serologic typing or higher resolution) and -DRB1 (at high resolution using DNA based typing). A 7/8 related donor match is permitted only if an 8/8 unrelated donor cannot be identified.
   2. Unrelated donor: must be a 7/8 or 8/8 match at HLA-A, -B, -C, and -DRB1 (at high resolution using DNA based typing).
6. Patients with adequate organ function as measured by:

   1. Cardiac: Left ventricular ejection fraction at rest ≥ 40% demonstrated by Multi Gated Acquisition Scan (MUGA) or echocardiogram. Patients with known heart disease must have a functional status no worse than American Heart Association Class I defined as patients with cardiac disease but without resulting limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea, or anginal pain.
   2. Hepatic:

   i. Total Bilirubin < 2.0 mg/dL (except for isolated hyperbilirubinemia attributed to Gilbert syndrome or antiretroviral therapy as specified in Appendix E) and alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 5x the upper limit of normal.

   ii. Concomitant Hepatitis: Patients with chronic hepatitis B or C may be enrolled on the trial providing the above bilirubin and transaminase criteria are met. In addition, there must be no clinical or pathologic evidence of irreversible chronic liver disease, and there must be no active viral replication as evidenced by an undetectable hepatitis viral load by a PCR-based assay.

   c) Renal: Creatinine clearance (calculated creatinine clearance is permitted) > 40 mL/min.

   d) Pulmonary: Diffusing capacity of the lung for carbon monoxide (DLCO), forced expiratory volume in one second (FEV1), or forced vital capacity (FVC) ≥ 45% of predicted (corrected for hemoglobin).
7. Signed Informed Consent

Exclusion Criteria:

1. Karnofsky/Lansky performance score < 70%.
2. Active central nervous system (CNS) malignancy; however, patients with a history of positive Cerebrospinal fluid (CSF) cytology that has become negative with intrathecal chemotherapy are eligible.
3. Uncontrolled bacterial, viral or fungal infection (currently taking medication and with progression or no clinical improvement).
4. Active Cytomegalovirus (CMV) retinitis or other CMV-related organ dysfunction.
5. AIDS related syndromes or symptoms that pose a perceived excessive risk for transplantation-related morbidity as determined by the principal investigator.
6. Untreatable HIV infection due to multidrug antiretroviral resistance. Patients with a detectable viral load > 750 copies/ml should be evaluated with an HIV drug resistance test (HIV-1 genotype). The results should be included as part of the Antiretroviral Review (described in Appendix D). This Review Committee will make the final determination as to whether HIV viremia could potentially be suppressed with alternate antiretroviral therapy. .
7. Pregnant (positive β-HCG) or breastfeeding.
8. Fertile men or women unwilling to use contraceptive techniques from the time of initiation of mobilization until six-months post-transplant.
9. Prior allogeneic HCT.
10. Patients with psychosocial conditions that would prevent study compliance and follow-up, as determined by the principal investigator.
11. T-cell depletion (including ATG or alemtuzumab) is not allowed.
12. Use of cord blood as the source of hematopoietic cells is not allowed.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Horowitz, MD, Study Director — Center for International Blood and Marrow Transplant Research
Locations (11):
- United States (11):
  - Mayo Clinic - Phoenix, Phoenix, Arizona
  - City of Hope National Medical Center, Duarte, California
  - University of CA, SF, San Francisco, California
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Blood & Marrow Transplant Program at Northside Hospital, Atlanta, Georgia
  - Johns Hopkins, Baltimore, Maryland
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - University of Texas/MD Anderson CRC, Houston, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in a manuscript and supporting information submitted to NIH BioLINCC (including data dictionaries, case report forms, data submission documentation, documentation for outcomes dataset, etc where indicated).
Supporting Information: Study Protocol, ICF
Time Frame: Within 6 months of official study closure at participating sites.
Access Criteria: Available to the public
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Result] Scott BL, Pasquini MC, Logan BR, Wu J, Devine SM, Porter DL, Maziarz RT, Warlick ED, Fernandez HF, Alyea EP, Hamadani M, Bashey A, Giralt S, Geller NL, Leifer E, Le-Rademacher J, Mendizabal AM, Horowitz MM, Deeg HJ, Horwitz ME. Myeloablative Versus Reduced-Intensity Hematopoietic Cell Transplantation for Acute Myeloid Leukemia and Myelodysplastic Syndromes. J Clin Oncol. 2017 Apr 10;35(11):1154-1161. doi: 10.1200/JCO.2016.70.7091. Epub 2017 Feb 13. PMID 28380315
- [Derived] Ambinder RF, Wu J, Logan B, Durand CM, Shields R, Popat UR, Little RF, McMahon DK, Cyktor J, Mellors JW, Ayala E, Kaplan LD, Noy A, Jones RJ, Howard A, Forman SJ, Porter D, Arce-Lara C, Shaughnessy P, Sproat L, Hashmi SK, Mendizabal AM, Horowitz MM, Navarro WH, Alvarnas JC. Allogeneic Hematopoietic Cell Transplant for HIV Patients with Hematologic Malignancies: The BMT CTN-0903/AMC-080 Trial. Biol Blood Marrow Transplant. 2019 Nov;25(11):2160-2166. doi: 10.1016/j.bbmt.2019.06.033. Epub 2019 Jul 4. PMID 31279752

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Allogeneic Transplant
Started | 20
Completed | 17
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: Transplanted participants
Arm/Group | Allogeneic Transplant
Number analyzed (Participants) | 17
Age, Continuous [Median (Full Range); unit: years] | 47 [25 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 11
  More than one race | 0
  Unknown or Not Reported | 2
Karnofsky Performance Score [Count of Participants; unit: Participants] — Assesses patient self-perceived global quality of life and functioning, where 100 equals perfect quality of life.
  Participants
    100 | 4
    90 | 9
    80 | 3
    70 | 1
Primary Malignancy [Count of Participants; unit: Participants]
  Acute Myeloid Leukemia (AML) | 9
  Acute Lymphocytic Leukemia (ALL) | 2
  Myelodysplastic Syndromes (MDS) | 2
  Hodgkin's Lymphoma | 1
  Non-Hodgkin's Lymphoma | 3
Leukemia Stage [Count of Participants; unit: Participants] — Population: Participants with leukemia (AML or ALL)
  Participants
    number analyzed (Participants) | 11
    First Complete Remission | 8
    Second Complete Remission | 3
Lymphoma Stage [Count of Participants; unit: Participants] — Population: Participants with lymphoma (Hodgkin's or non-Hodgkin's)
  Participants
    number analyzed (Participants) | 4
    Complete Remission | 3
    Partial Remission | 1
HIV Viral Load [Count of Participants; unit: Participants]
  Undetectable by Assay | 15
  Detectable by Assay | 2
Recipient Cytomegalovirus Status [Count of Participants; unit: Participants]
  Positive | 12
  Negative | 5
Number of Regimens of Induction Chemotherapy [Count of Participants; unit: Participants]
  1 | 10
  2 | 6
  3 | 1
Number of Regimens of Salvage Chemotherapy [Count of Participants; unit: Participants]
  0 | 10
  1 | 6
  3 | 1
Donor Type [Count of Participants; unit: Participants] — Donor/recipient matching described by relatedness and HLA matching. A matched donor corresponds to matching on 8/8 HLA loci, while mismatched donor indicates 7/8 matching.
  Participants
    Matched Related | 4
    Matched Unrelated | 9
    Mismatched Related | 3
    Mismatched Unrelated | 1
CD4 T-cell Count [Median (Full Range); unit: cells/microliter] | 224 [55 to 833]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Non-Relapse Mortality
Description: The events for non-relapse mortality are death due to any cause other than relapse of the underlying malignancy.
Time Frame: Day 100, 1 Year, and 2 Years Post-transplant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Allogeneic Transplant
Number analyzed (Participants) | 17
percentage of participants
  Day 100 | 0.0 [0.0 to 0.0]
  1 Year | 11.8 [1.8 to 32.2]
  2 Years | 18.3 [4.1 to 40.7]

2. Secondary Outcome: Percentage of Participants With Overall Survival
Description: Overall survival is defined as the time from transplant to death from any cause.
Time Frame: Six months, 1 Year, and 2 Years Post-transplant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Allogeneic Transplant
Number analyzed (Participants) | 17
percentage of participants
  6 Months | 82.4 [54.7 to 93.9]
  1 Year | 58.8 [32.5 to 77.8]
  2 Years | 50.2 [24.3 to 71.4]

3. Secondary Outcome: Percentage of Participants With Relapse/Progression
Description: Relapse/Progression is defined as relapse or progression of the primary malignancy.
Time Frame: 1 Year Post-transplant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Allogeneic Transplant
Number analyzed (Participants) | 17
percentage of participants | 29.4 [10.2 to 51.9]

4. Secondary Outcome: Primary Cause of Death
Time Frame: Up to 2 Years Post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic Transplant
Number analyzed (Participants) | 17
Participants
  Relapse/Progresion | 5
  Acute GVHD | 1
  Adult Respiratory Distress Syndrome | 1
  Liver Failure | 1
  Still Alive | 9

5. Secondary Outcome: Disease Status
Description: Patients will be assessed for disease status at Day 100 post-HCT, classified as complete remission, partial remission, stable disease, and relapse/progressive disease.
Time Frame: Day 100 Post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic Transplant
Number analyzed (Participants) | 17
Participants
  Complete remission | 13
  Relapse/progressive disease | 4

6. Secondary Outcome: Percentage of Participants Recovering Hematologic Function
Description: Recovery of hematologic function is described by the time to neutrophil and platelet recovery. Time to neutrophil recovery will be the first of three consecutive days of > 500 neutrophils/μL following the expected nadir. Time to platelet engraftment will be described by the date when platelet count is > 20,000/μL for the first of three consecutive labs with no platelet transfusions 7 days prior.
Time Frame: Days 28 and 100 Post-transplant
Measure: Number; unit: percentage of participants
Arm/Group | Allogeneic Transplant
Number analyzed (Participants) | 17
percentage of participants
  Day 28 Neutrophil Recovery | 100.0
  Day 100 Platelet Recovery | 94.1

7. Secondary Outcome: Chimerism
Description: Donor T-cell and myeloid chimerism will be described separately by conditioning regimen intensity (myeloablative or reduced intensity) according to proportions with mixed chimerism (5-95% donor cells out of all), full chimerism (>95% donor cells), or graft rejection (<5% donor cells).
Time Frame: Week 4, Day 100, and 6 months Post-transplant
Measure: Count of Participants; unit: Participants
Groups:
- Myeloablative Allogeneic Transplant: Myeloablative conditioning (MAC) (Busulfan and Fludarabine or Cyclophosphamide and Total Body Irradiation) will be administered prior to allogeneic hematopoietic cell transplantation (HCT).
- Reduced Intensity Allogeneic Transplant: Reduced-intensity conditioning (RIC) (Fludarabine and Busulfan; or Fludarabine and Melphalan) will be administered prior to allogeneic hematopoietic cell transplantation (HCT).
Arm/Group | Myeloablative Allogeneic Transplant | Reduced Intensity Allogeneic Transplant
Number analyzed (Participants) | 8 | 9
Participants
  Week 4: Full Chimerism | 4 | 5
  Week 4: Mixed Chimerism | 2 | 4
  Week 4: Graft Rejection | 1 | 0
  Week 4: Dead at Assessment | 0 | 0
  Week 4: No Assay Reported | 1 | 0
  Day 100: Full Chimerism | 3 | 5
  Day 100: Mixed Chimerism | 4 | 4
  Day 100: Graft Rejection | 0 | 0
  Day 100: Dead at Assessment | 1 | 0
  Day 100: No Assay Reported | 0 | 0
  6 Months: Full Chimerism | 4 | 5
  6 Months: Mixed Chimerism | 2 | 2
  6 Months: Graft Rejection | 0 | 0
  6 Months: Dead at Assessment | 2 | 2
  6 Months: No Assay Reported | 0 | 0

8. Secondary Outcome: Percentage of Participants With Acute Graft-Versus-Host Disease (GVHD)
Description: Acute GVHD is graded according to the scoring system proposed by Przepiorka et al.1995:
  Skin stage:
  0: No rash
  1. Rash <25% of body surface area
  2. Rash on 25-50% of body surface area
  3. Rash on > 50% of body surface area
  4. Generalized erythroderma with bullous formation
  Liver stage (based on bilirubin level)*:
  0: <2 mg/dL 1.2-3 mg/dL 2.3.01-6 mg/dL 3.6.01-15.0 mg/dL 4.>15 mg/dL
  GI stage*:
  0: No diarrhea or diarrhea <500 mL/day
  1. Diarrhea 500-999 mL/day or persistent nausea with histologic evidence of GVHD
  2. Diarrhea 1000-1499 mL/day
  3. Diarrhea >1500 mL/day
  4. Severe abdominal pain with or without ileus * If multiple etiologies are listed for liver or GI, the organ system is downstaged by 1.
  GVHD grade:
  0: All organ stages 0 or GVHD not listed as an etiology I: Skin stage 1-2 and liver and GI stage 0 II: Skin stage 3 or liver or GI stage 1 III: Liver stage 2-3 or GI stage 2-4 IV: Skin or liver stage 4
Time Frame: Day 100 Post-transplant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Allogeneic Transplant
Number analyzed (Participants) | 17
percentage of participants
  Grade II-IV Acute GVHD | 41.2 [17.8 to 63.4]
  Grade III-IV Acute GVHD | 11.8 [1.8 to 31.9]

9. Secondary Outcome: Percentage of Participants With Chronic Graft-Versus-Host Disease (GVHD)
Description: Chronic GVHD is classified per 2005 NIH Consensus Criteria (Filipovich et al. 2005) into categories of severity: none, mild, moderate, and severe. Occurrence of chronic GVHD is defined as the occurrence of mild, moderate, or severe chronic GVHD per this classification.
Time Frame: 1 Year Post-transplant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Allogeneic Transplant
Number analyzed (Participants) | 17
percentage of participants | 17.6 [4.0 to 39.2]

10. Secondary Outcome: Infection Severity
Description: The maximum grade of infections reported by participants are described, as defined in the BMT CTN Technical MOP.
Time Frame: 1 Year Post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic Transplant
Number analyzed (Participants) | 17
Participants
  Grade 0-1 | 6
  Grade 2 | 3
  Grade 3 | 8

ADVERSE EVENTS:
Time Frame: Up to 2 Years Post-transplant
Arm/Group | Allogeneic Transplant
All-Cause Mortality (participants affected / at risk) | 8/20
Serious Adverse Events (participants affected / at risk) | 5/20
Other Adverse Events (participants affected / at risk) | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allogeneic Transplant (N=20)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (3)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2014-02-18): https://cdn.clinicaltrials.gov/large-docs/44/NCT01410344/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2018-03-23): https://cdn.clinicaltrials.gov/large-docs/44/NCT01410344/SAP_001.pdf